CLINICAL TRIAL: NCT00137917
Title: A Primary Vaccination Study to Evaluate Immunogenicity, Safety and Reactogenicity of 3 Doses of GSK Biologicals/Finlay's Meningococcal B Candidate Vaccine Given Intramuscularly Using Either 0-2-4 Month or 0-1-6 Month Schedule to Healthy Subjects Aged 12-18 Years
Brief Title: Immunogenicity & Safety Study of a Meningococcal Serogroup B Vaccine Given in a 3 Dose Schedule to Healthy Adolescents Aged 12-18 Yrs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 710158/002
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
Keywords: Prophylaxis meningococcal serogroup B disease
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

INTERVENTIONS:
Biological: Meningococcal serogroup B vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of 3 doses of the meningococcal serogroup B vaccine when given, using either a 0-2-4 month or a 0-1-6 month schedule, to healthy adolescents aged 12-18 years; a control group will receive 2 doses of Havrix™ (0-6 months) and Meningitec™ (month 1).

DETAILED DESCRIPTION:
The study is open; however, vaccines given to study group at 0-1-6 months and to control group will be administered in an observer-blind manner. 3 blood samplings for antibody testing: before vaccination and one month after the second and third vaccine doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between, and including, 12 and 18 years of age at the time of the first vaccination.
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Previous vaccination against or history of meningococcal B or C, or hepatitis A disease or exposure to meningococcal B disease within last year.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 478 (Actual)
Dates: Start 2002-07; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Meningococcal serogroup B (MenB) immune response (i.e. at least a 4-fold increase in serum bactericidal activity [SBA] from pre-vaccination titer) at 1 month postvaccination for each MenB strain assayed

SECONDARY OUTCOMES:
For each MenB strain assayed, pre and 1m post dose 2 and 3: SBA seropositivity, titer and immune response (post dose 2 only)
After each vaccination: grade 3 and any solicited symptoms (Day 0-14), unsolicited symptoms (Day 0-30)
Serious adverse events [SAEs] (whole study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Boutriau D, Poolman J, Borrow R, Findlow J, Domingo JD, Puig-Barbera J, Baldo JM, Planelles V, Jubert A, Colomer J, Gil A, Levie K, Kervyn AD, Weynants V, Dominguez F, Barbera R, Sotolongo F. Immunogenicity and safety of three doses of a bivalent (B:4:p1.19,15 and B:4:p1.7-2,4) meningococcal outer membrane vesicle vaccine in healthy adolescents. Clin Vaccine Immunol. 2007 Jan;14(1):65-73. doi: 10.1128/CVI.00230-06. Epub 2006 Oct 25. PMID 17065257
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 710158/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 710158/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 710158/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 710158/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 710158/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register